CLINICAL TRIAL: NCT02974894
Title: The Effects of Lactobacillus Plantarum on Cortisol, IgA and Alpha-amylase Levels in Human Saliva During Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Exjobb stress
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Stress Reaction
MeSH Terms: conditions — Fractures, Stress | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Capsules containing potato starch as a filler and Lactobacillus plantarum
  Interventions: Dietary Supplement: Probiotic (Lactobacillus Plantarum)
- Placebo (Placebo Comparator): Capsules containing potato starch
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic (Lactobacillus Plantarum)
  Arms: Probiotic
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
In the present study the main goal has been to clarify the effect of the probiotic bacteria Lactobacillus plantarum 299v on the salivary cortisol level in young adults under examination stress. Salivary IgA from minor glands and in whole human saliva was measured as alternative marker of stress. The hypothesis was that the levels of cortisol would be reduced or stabilized in the test group in comparison to the placebo group where the cortisol levels were expected to increase due to the examination-induced stress. By contrast, the salivary IgA levels were expected to increase in the test group in comparison to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* adults
* studying at the University in Lund
* participation in ongoing examination period

Exclusion Criteria:

* pregnancy
* intake of antibiotics
* medication with cortisone during the study period

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The impact of Lactobacillus plantarum on the levels of stress-induced cortisol in saliva. | Change from baseline in cortisol levels at 14 days

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersson H, Tullberg C, Ahrne S, Hamberg K, Lazou Ahren I, Molin G, Sonesson M, Hakansson A. Oral Administration of Lactobacillus plantarum 299v Reduces Cortisol Levels in Human Saliva during Examination Induced Stress: A Randomized, Double-Blind Controlled Trial. Int J Microbiol. 2016;2016:8469018. doi: 10.1155/2016/8469018. Epub 2016 Dec 22. PMID 28101105